CLINICAL TRIAL: NCT07049744
Title: Bilateral Hypoglossal Nerve Stimulation With the XII Medical HGNS System for the Treatment of Adult Obstructive Sleep Apnea Pilot Study
Brief Title: Hypoglossal Nerve Stimulation for the Treatment of Adult Obstructive Sleep Apnea
Acronym: BEAT OSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: XII Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: XII-002
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: OSA; HGNS
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- XII Medical HGNS System (Experimental): Participants receiving HGNS using the XII Medical System
  Interventions: Device: XII Medical HGNS System

INTERVENTIONS:
Device: XII Medical HGNS System — XII Medical HGNS System

SUMMARY:
The goal of this interventional study is to assess the safety and performance of the XII Medical Hypoglossal Nerve Stimulation (HGNS) System in people who have moderate to severe Obstructive Sleep Apnea (OSA).

Participation in this study involves being implanted with a Neurostimulator which provides electrical stimulation of the hypoglossal nerve (HGN). Participants will receive treatment at home during sleep, and participate in sleep studies to track and record the quality of the sleep. Participants will be monitored over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≤ 32 kg/m2
* AHI of 15-50 events/hour
* Central + mixed apnea index ≤ 25%
* Participants who have either not tolerated, have failed or refused positive airway pressure (PAP)

Exclusion Criteria:

* Pregnancy or breast-feeding.
* Significant upper airway anatomic abnormalities
* Hypoglossal nerve weakness
* Central sleep apnoea condition
* Significant positionally-dependent OSA.
* Complete concentric patterns of soft palate collapse on DISE
* Inadequately treated non-OSA sleep disorder(s).
* Significant co-morbidities or prior surgeries that contra-indicate a surgical procedure or general anesthesia
* Taking medications that in the opinion of the investigator may alter consciousness, the pattern of respiration, or sleep architecture
* Participants on a GLP-1

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Safety of the XII Medical HGNS System | Six months post-implantation
  Assessment of serious adverse device events

SECONDARY OUTCOMES:
Performance of the XII Medical HGNS System | Six months post-implantation
  Change from baseline and Responder Rates for the Apnea Hypopnea Index
Performance of the XII Medical HGNS System | Six months post-implantation
  Change from baseline and Responder Rates for the Oxygen Desaturation Index

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Canberra ENT, Canberra, Australian Capital Territory
  - Westmead Hospital / Chris O'Brien Lifehouse, Sydney, New South Wales
  - The Wollongong Hospital, Wollongong, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Perth Head & Neck Surgery, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No